CLINICAL TRIAL: NCT07200869
Title: Vaso-occlusive Crisis Incidence and Outcomes in a Pediatric Sickle Cell Population
Brief Title: Outcomes of Vaso-occlusive Crisis in Pediatric Sickle Cell Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nadia Fawzy Fahmy Hanna, Principle investigator, Assiut University
Other Study IDs: Pediatric sickle cell crises
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis
Keywords: Pediatric; Sickle Cell Anemia; Incidence; Outcomes
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle Cell pediatric patients: Children with sickle cell disease whose medical records will be retrospectively reviewed at Assiut University Hospital.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — retrospective observational study. No intervention will be administered; data will be collected from existing medical records of pediatric sickle cell patients at Assiut University Hospital.

SUMMARY:
This study aims to assess the incidence and clinical outcomes of vaso-occlusive crises in pediatric patients with sickle cell disease. Data will be collected and analyzed to identify risk factors and related complications.

DETAILED DESCRIPTION:
Sickle cell disease is a hereditary blood disorder characterized by the presence of sickle-shaped red blood cells, which leads to recurrent vaso-occlusive crises (VOC). These painful episodes are among the most common causes of hospitalization and are associated with significant morbidity in pediatric patients. Despite ongoing improvements in the management of sickle cell disease, there is still limited data describing the incidence, risk factors, and clinical outcomes of VOC in children within our population.

This study is designed to retrospectively analyze medical records of pediatric patients with sickle cell disease at Faculty of Medicine, Assiut University. The primary aim is to estimate the incidence of vaso-occlusive crises and to identify the most frequent complications. Secondary objectives include evaluating treatment approaches, length of hospital stay, and clinical outcomes. Findings from this study are expected to provide valuable insights that may help improve clinical care strategies and preventive measures for affected children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-18 years. Confirmed diagnosis of sickle cell anemia by hemoglobin electrophoresis or high-performance liquid chromatography .

History of at least one hospital visit or admission for vaso-occlusive crisis

Exclusion Criteria:

* Patients with other hemoglobinopathies (e.g., thalassemia). Patients with incomplete medical records. Children with coexisting chronic diseases that may confound pain crises .

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients (1-18 years) with confirmed Sickle Cell Disease. The study observes the incidence and outcomes of vaso-occlusive crises (VOCs). Both sexes are eligible. Healthy volunteers are not included.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of vaso-occlusive crisis in pediatric sickle cell patients | Retrospective review of medical records from 2019 to 2024
  Frequency of vaso-occlusive crisis episodes will be identified through retrospective chart review of pediatric sickle cell patients.

SECONDARY OUTCOMES:
Complications associated with vaso-occlusive crisis (e.g., acute chest syndrome, stroke, infections) | Throughout the study period (2019-2024)
  Complications related to vaso-occlusive crisis will be identified and documented from patient records.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vichinsky EP, Neumayr LD, Earles AN, Williams R, Lennette ET, Dean D, Nickerson B, Orringer E, McKie V, Bellevue R, Daeschner C, Manci EA. Causes and outcomes of the acute chest syndrome in sickle cell disease. National Acute Chest Syndrome Study Group. N Engl J Med. 2000 Jun 22;342(25):1855-65. doi: 10.1056/NEJM200006223422502. PMID 10861320
- [Background] Powars DR, Chan LS, Hiti A, Ramicone E, Johnson C. Outcome of sickle cell anemia: a 4-decade observational study of 1056 patients. Medicine (Baltimore). 2005 Nov;84(6):363-376. doi: 10.1097/01.md.0000189089.45003.52. PMID 16267411
- [Background] Platt OS, Thorington BD, Brambilla DJ, Milner PF, Rosse WF, Vichinsky E, Kinney TR. Pain in sickle cell disease. Rates and risk factors. N Engl J Med. 1991 Jul 4;325(1):11-6. doi: 10.1056/NEJM199107043250103. PMID 1710777
- [Background] Serjeant GR. The natural history of sickle cell disease. Cold Spring Harb Perspect Med. 2013 Oct 1;3(10):a011783. doi: 10.1101/cshperspect.a011783. PMID 23813607
- [Background] El-Beshlawy A, Youssry I. Prevention of hemoglobinopathies in Egypt. Hemoglobin. 2009;33 Suppl 1:S14-20. doi: 10.3109/03630260903346395. PMID 20001619
- [Background] Piel FB, Hay SI, Gupta S, Weatherall DJ, Williams TN. Global burden of sickle cell anaemia in children under five, 2010-2050: modelling based on demographics, excess mortality, and interventions. PLoS Med. 2013;10(7):e1001484. doi: 10.1371/journal.pmed.1001484. Epub 2013 Jul 16. PMID 23874164
- [Background] Rees DC, Williams TN, Gladwin MT. Sickle-cell disease. Lancet. 2010 Dec 11;376(9757):2018-31. doi: 10.1016/S0140-6736(10)61029-X. Epub 2010 Dec 3. PMID 21131035